CLINICAL TRIAL: NCT05956132
Title: Retrospective Analysis of Clinical and Biochemical Features for the Identification of Dominant Inheritance of Calpainopathies
Brief Title: Clinical and Biochemical Features for the Identification of Dominant Calpainopathies
Acronym: DOM-CAL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other); Istituto Giannina Gaslini (Other); Ospedale Policlinico San Martino (Other); Universita di Verona (Other); Azienda Ospedaliera Universitaria Senese (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.08
Record Dates: First submitted 2023-06-30; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Calpain-3 Deficiency Limb Girdle Muscular Dystrophy Type 2A
MeSH Terms: conditions — Limb-girdle muscular dystrophy type 2A | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective study — data collection from clinical history and medical records

SUMMARY:
Mutations in the CAPN3 gene cause muscular dystrophies with dysfunction in calpain-3. Calpainopathies are usually inherited in an autosomal recessive manner but in some families they can occur in a dominant inheritance. The significance of heterozygous variants is difficult to interpret in the absence of family history. In this study, the investigators will review the clinical and laboratory information in a cohort of patients identified in the participating centers, with the aim of improving the diagnostic strategy of dominant calpainopathies.

DETAILED DESCRIPTION:
The investigators will review clinical and biomarker information in a cohort of 50 patients with heterozygous variants in the CAPN3 gene. Patients are referred by participating centers who will provide anonymised information on the clinical phenotype and laboratory test results. Suitable subjects will be contacted to obtain informed consent. Pseudonymised anamnestic data will be collected from the patient's clinical history and medical records.The aim is to identify a set of multidisciplinary data sufficient to define a diagnostic algorithm for the dominant calpainopathies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical LGMD phenotype, family history with dominant inheritance or sporadic cases, single variant in CAPN3, second variant excluded by MLPA (Multiplex Ligation Probe Amplification) or by analysis of mRNA extracted from muscle.

Exclusion Criteria:

* No variants in CAPN3, two variants in CAPN3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Suitable subjects identified in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Muscle strenght | through study completion, an average of 1 year
  Evaluation of muscle strength with MRC Scale (score 1-5 from weaker to stronger)
Muscle biopsy | through study completion, an average of 1 year
  Evaluation of histology and calpain 3 expression (present, reduced, absent)
Creatin Kinase | through study completion, an average of 1 year
  Amount of creatine kinase in blood in units (U) of enzyme activity per liter (L) of serum
Clinical history | through study completion, an average of 1 year
  Data collection sheet from clinical records

CONTACTS AND LOCATIONS:
Overall Officials: RITA BARRESI, DR, Principal Investigator — IRCCS SAN CAMILLO
Locations (2):
- Italy (2):
  - San Camillo Irccs, Venice-Lido, VE
  - IRCCS San Camillo, Venice-Lido

IPD SHARING:
Plan to Share IPD: No
Data and images may be disclosed in strictly anonymous form through meetings, conferences and scientific publications. In any case, the name or any other detail suitable for identifying the individual participant will not be disclosed as the data may only be presented in aggregate form.

REFERENCES:
- [Derived] D'Este G, Giorgetti A, Cassandrini D, Magri F, Ronchi D, Rubegni A, Lopergolo D, Malandrini A, Merlini L, Vattemi G, Tonin P, Barresi R. Recurrent CAPN3 p.Asp753Asn Variant Supports a Potential Dominant Calpainopathy with Variable Clinical Expressivity. Int J Mol Sci. 2025 Nov 25;26(23):11384. doi: 10.3390/ijms262311384. PMID 41373542